CLINICAL TRIAL: NCT05700773
Title: Assessing the Relationship Between Myonectin Concentration and the Course of Hospitalization and the 30-day Risk of Cardiac Endpoints in Patients With the First Incident of ST-segment Elevation Mycardial Infarction Treated With Primary PCI
Brief Title: The Relationship Between Myonectin Concentration and the Course of ST-segment Elevation Myocardial Infarction
Status: Recruiting | Type: Observational
Sponsor: Michał Jaśkiewicz (Other)
Collaborators: Jan Biziel University Hospital No 2 in Bydgoszcz (Other)
Responsible Party: Sponsor-Investigator, Michał Jaśkiewicz, Principal Investigator; Consultant in Interventional Cardiology, Wojewodzki Szpital Zespolony w Elblagu
Organization: Wojewodzki Szpital Zespolony w Elblagu (Other)
Other Study IDs: wszz0001
Record Dates: First submitted 2022-12-26; First posted 2023-01-26 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: ST Elevation Myocardial Infarction
Keywords: myonectin; CTRP15; primary percutaneous coronary intervention; troponin concentration; ejection fraction; echocardiography; 30-day mortality; One-year mortality; Physical Activity Questionnaire Short Form; skeletal muscle mass
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to test the potentially protective role of myonectin in patients with a first episode of ST elevation myocardial infarction (MI) treated with primary percutaneous coronary intervention (PCI).

The main questions which are assumed to be answered after study completion:

1. Does higher myonectin concentration influence the in-hospital and 30-day course of the first ST-elevation MI in patients treated with primary coronary angioplasty
2. Is there a relationship between the serum myonectin concentration, related to patient's nutritional status and physical activity with the patient's physical activity declared as usually before the coronary event occurrence, the cardiac biomarkers level, and myocardial and skeletal muscle mass determined in order to objectify the relationship of physical activity before the infarction with 30-day and one-year mortality, and the other primary and secondary outcomes measured at 12-month visit, e.g. the extent of myocardial infarction,
3. Is there a relationship between the baseline concentration of myonectin and troponin with the control of atherosclerosis risk factors, declared physical activity and parameters of body composition, outcome of treadmill exercise test, values of echocardiographic parameters and myonectin concentration 12 months after a cardiovascular incident

DETAILED DESCRIPTION:
Myonectin or Complement C1q Tumor Necrosis Factor - Related Protein 15 (CTRP15) is a cytokine secreted by skeletal muscle. The participation of myonectin in the regulation of lipid homeostasis in the liver and adipose tissue has been proven. The concentration of myonectin depends on the nutritional status of the organism, it decreases during fasting and increases after feeding. In studies on mice, a protective effect of high concentrations of myonectin on the course of myocardial infarction was observed. The effect of regular physical exercise on the concentration of myonectin in the serum was also demonstrated. Abnormal function of myokines, including myonectin, has also been linked to sarcopenia, which significantly negatively affects the prognosis of patients with heart failure.

Potentially protective properties of myonectin in the case of ischemia-reperfusion injury in the course of myocardial infarction have not been studied in humans so far.

Myonectin may become a potentially useful prognostic indicator of the severity of myocardial infarction. It may also potentially become a target for a new cardioprotective therapy in patients with acute myocardial ischaemia.

ELIGIBILITY:
Inclusion Criteria:

* symptoms of acute coronary syndrome
* acute ST segment elevation in two or more leads in ECG
* primary PCI

Exclusion Criteria:

* pregnancy
* patients unconscious, with altered consciousness or not able to cooperate
* cardiogenic shock
* significant physical effort within 24 hours before onset of MI
* active infection at admission, intramuscular injection
* myocardial infarction in patient's medical history
* heart failure New York Heart Association (NYHA) class III - IV in patient's medical history
* renal failure (chronic kidney disease, CKD) with glomerular filtration rate (GFR) < 30ml/min
* history of malignant neoplasms in the last 5 years
* patients incapacitated, active soldiers, imprisoned or related with investigators

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the study site with a diagnosis of STEMI treated with primary PCI who consent to follow-up during the scheduled enrollment window.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
30-day mortality | 30 days
  All-cause mortality
12-month mortality | 12 months
  All-cause mortality
Myocardial infarction | 12 months
  Any myocardial infarction during follow-up
Stroke | 12 months
  Any stroke or transient ischaemic attack (TIA) during follow-up
Bleeding | 12 months
  Any registered clinically significant bleeding

SECONDARY OUTCOMES:
Left Ventricular Ejection Fraction | up to 7 days and 12 months
  Left Ventricular Ejection Fraction in echocardiography, the absolute value and change after 12 months
Cardiac Troponin T | up to 7 days
  Highest registered concentration of high sensitive Cardiac Troponin T during hospitalization
Left Ventricular Internal Dimension at End of Diastole (LVIDd) | up to 7 days and 12 months
  Left Ventricular Internal Dimension at End of Diastole (LVIDd) in echocardiography, the absolute value and change after 12 months
Length of hospitalization | 30 days
  Length of in-hospital stay (LOS)
Myonectin serum concentration | up to 7 days and 12 months
  Change of myonectin concentration after 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michał Jaśkiewicz, MD, Principal Investigator — Voivodeship Hospital in Elblag, Poland; Department of Cardiology; Jacek Budzyński, MD PhD, Principal Investigator — Jan Biziel University Hospital No 2 in Bydgoszcz, Poland; Department of Vascular and Internal Diseases, Nicolaus Copernicus University in Torun, Collegium Medicum in Bydgoszcz, Poland
Locations (1):
- Voivodeship Hospital in Elblag, Elblag, Warmian-Masurian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided